CLINICAL TRIAL: NCT07087327
Title: A Phase 3, Multicenter, Open-label, Uncontrolled, Long-term Japan-China Joint Trial to Evaluate the Safety and Efficacy of EB-1020 QD XR Capsules Administered Orally Once Daily in Children and Adolescents With Attention- Deficit/Hyperactivity Disorder
Brief Title: A Long-term Trial of EB-1020 in Pediatric Patients With ADHD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 405-102-00115
Record Dates: First submitted 2025-07-24; First posted 2025-07-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Attention-Deficit Hyperactivity Disorder(ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EB-1020 (QD XR Capsules) low dose (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) low dose
- EB-1020 (QD XR Capsules) high dose (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) high dose

INTERVENTIONS:
Drug: EB-1020 (Centanafadine) low dose — low dose, capsule, oral, once daily, for 52 weeks
  Arms: EB-1020 (QD XR Capsules) low dose
Drug: EB-1020 (Centanafadine) high dose — high dose, capsule, oral, once daily, for 52 weeks
  Arms: EB-1020 (QD XR Capsules) high dose

SUMMARY:
The purpose of this study is to evaluate the safety of long-term administration of mainly high doses of EB-1020 over 52 weeks in pediatric ADHD patients.

ELIGIBILITY:
Inclusion Criteria:

<Rollover participants>

* Participants who completed the 6-week treatment period and 1-week follow-up period in the preceding double-blind parent trial and did not meet the criteria for discontinuation of the IMP at Week 6.
* Participants who have not been found to have major problems with trial requirements, such as compliance with the IMP, in the preceding double-blind parent trial.

<De novo participants>

* Participants with a primary diagnosis of ADHD based on DSM-5 diagnostic criteria, differentiated from other mental disorders using the MINI-KID, excluding other specified ADHD or unspecified ADHD.
* Participants with a symptom total raw score of >= 28 on the ADHD-RS-5 at baseline.
* Participants with a score of 4 or higher on the Clinical Global Impression Severity - ADHD (CGI-S-ADHD) at baseline.

Exclusion Criteria:

<Rollover participants>

* Participants who have a positive pregnancy test result at baseline.
* Participants who were found to have serious or severe adverse events that were judged to be related to the IMP in the preceding double-blind parent trial.
* Participants who have a significant risk of committing suicide in the opinion of the investigator or subinvestigator, or based on the following evidence.

  * Active suicidal ideation as evidenced by an answer of "yes" on Questions 4 or 5 on the section of suicidal ideation or reported suicidal behavior on the since last visit version of the Columbia-Suicide Severity Rating Scale (C SSRS) in the preceding double-blind parent trial.
* Participants who plan to use prohibited medication during the trial. Participants who used prohibited medication during the preceding double-blind parent trial should be excluded if the investigator or subinvestigator judges that there is a possibility of repeated use of prohibited medication.

<De novo participants>

* Participants who have a positive pregnancy test result at baseline.
* Participants determined to have the following diseases based on an interview using the MINI-KID.

  * Tourette's disorder
  * Panic disorder
  * Conduct disorder
  * Psychotic disorder
  * Post-traumatic stress disorder
  * Bipolar disorder
* Participants with a generalized anxiety disorder requiring pharmacotherapy, based on the DSM-5 diagnostic criteria.
* Participants with an autism spectrum disorder based on the DSM-5 diagnostic criteria.
* Participants with a personality disorder, oppositional defiant disorder, or obsessive-compulsive disorder that is the primary focus of treatment, based on the DSM-5 diagnostic criteria.
* Participants with a diagnosis of major depressive disorder (MDD), based on the DSM-5 diagnostic criteria who currently have a major depressive episode, or who have required treatment for MDD within the past 3 months prior to screening. Also, participants who, in the judgment of the investigator or subinvestigator, may have a worsening of MDD during the trial or may require treatment during the trial period.
* Participants who have a diagnosis of intellectual disability with an intelligence quotient (IQ) score less than 70.
* Participants who have a significant risk of committing suicide in the opinion of the investigator or subinvestigator, or based on the following evidence.

  * Active suicidal ideation as evidenced by an answer of "yes" on Questions 4 or 5 (over the last 6 months) on the section of suicidal ideation or a history of suicidal behavior (over the last 6 months) on the Baseline/Screening version of the C-SSRS at screening.
* Participants with a diagnosis of substance use disorder.
* Participants who have laboratory test results at screening as follows:

  * Platelets<=130,000/mm3
  * Hemoglobin<=11.2 g/dL
  * Neutrophils, absolute<=1000/mm3
  * AST > 2 x ULN
  * ALT > 2 x ULN
  * eGFR < 45 mL/min/1.73 m2, calculated by the CKiD U25 equation
  * CPK>=2 x ULN (except for the participants that the medical monitor determines that inclusion is possible based on discussion about their condition with the investigator or subinvestigator)
  * Abnormal values for both free T4 and TSH
* Participants who cannot agree to discontinuation of prohibited concomitant medication, such as ADHD medication or antidepressants.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Experiencing Treatment-Emergent Adverse Events (TEAEs) | Baseline, week52
  An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs with an onset date on or after the first dose of IMP. They are all adverse events that started after the start of centanafadine; or if the event was continuous from baseline and was worsening, serious, study drug-related, or resulted in death, discontinuation, interruption or reduction of study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Hokkaido University Hospital, Sapporo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.